CLINICAL TRIAL: NCT04751604
Title: Improvement of the Nutritional Status Regarding Nicotinamide (Vitamin B3) and the Disease Course of COVID-19
Acronym: COVit-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: A 107/20
Record Dates: First submitted 2021-02-03; First posted 2021-02-12 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide (Experimental): Daily oral administration of 1,000 mg nicotinamide [1x 500-mg conventional nicotinamide tablet and 1x 500-mg tablet with controlled-ileocolonic-release nicotinamide (CICR-NAM)] for 4 weeks
  Interventions: Dietary Supplement: Nicotinamide
- Placebo (Placebo Comparator): Daily oral administration of 2 matching placebo tablets for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide — Daily oral administration of 1,000 mg nicotinamide [1x 500-mg conventional nicotinamide tablet and 1x 500-mg tablet with controlled-ileocolonic-release nicotinamide (CICR-NAM)] for 4 weeks
  Arms: Nicotinamide
Dietary Supplement: Placebo — Daily oral administration of 2 matching placebo tablets for 4 weeks
  Arms: Placebo

SUMMARY:
Based on the literature, it seems likely that a nutritional intervention with nicotinamide (a form of vitamin B3) can support the therapy of SARS-CoV-2 infection (COVID-19). A pilot phase of the COVit trial showed an effect of nicotinamide on the time to complete resolution of COVID-19 symptoms. In addition, diarrhoea is a common symptom of COVID-19. Therefore, in a second part of the study, 420 symptomatic patients each with confirmed SARS-CoV-2 infection are to take 1,000 mg nicotinamide (500 mg conventional nicotinamide and 500 mg nicotinamide released in a controlled manner in the intestine) or corresponding placebos per day in a blinded fashion for 4 weeks. The primary endpoint of the trial is the occurrence of individual COVID-19 symptoms over time (primary analysis time point: week 2). Secondary endpoints focus on the severity of COVID-19 symptoms, the post-COVID-19 syndrome (PCS), anti-SARS-CoV-2 antibody levels, and the time to resolution of individual or all symptoms. Exploratory endpoints include the WHO clinical scale for COVID-19, development of severe COVID-19, fatigue, quality of life and biomarkers. Patients are approached after positive testing and give their informed consent online. After randomised distribution of the trial supplements, patients are interviewed by telephone about their disease course at baseline (week 0), week 2, week 4, week 6 and after 6 months. Stool samples are collected from up to 400 patients at the same timepoints. In addition to blood count and standard blood profile, various inflammatory markers and the metabolome, in particular tryptophan metabolism, are examined in the blood of up to 20 selected patients. In these patients, the viral strain is determined by sequencing from nasopharyngeal swabs. In selected patients, short-term pharmacokinetics of nicotinamide, nicotinic acid and nicotinuric acid as well as of metabolites of nicotinamide and tryptophan are investigated. In the stool, changes in the microbiome (in 100-300 patients) as well as metagenome and metabolome (in a subgroup) will be analysed. The study is expected to produce rapid results on whether nicotinamide supplementation can alleviate the disease course of COVID-19. Moreover, a follow-up interview, a smell test, a cognitive test and anti-SARS-CoV-2 antibody levels after at least 6 months will be used to investigate whether the supplementation has any influence on PCS as well as the immune reaction against SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* The patient is of age (at least 18 years).
* SARS-CoV-2 infection confirmed by laboratory findings; the positive test must not date back more than 7 days.
* Relevant infection symptoms, e.g. in the respiratory or gastrointestinal tract.
* The patient has been able to give written consent via a website before any trial procedure is performed and can comply with the trial-dependent prerequisites and requirements.

Exclusion Criteria:

* Current participation in another trial.
* Pregnancy or breastfeeding.
* Vaccination against SARS-CoV-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Frequencies of individual COVID-19 symptoms at week 0, week 2 (primary time of analysis), week 4 and week 6 as well as after 6 months. | Through study completion, up to 6 months
  A broad range of symptoms is recorded during telephone interviews at baseline, at weeks 2, 4 and 6 and after 6 months in an electronic case report form. Key symptoms include performance drop / limited physical capacity, the ability to perform normal activities, cough and fatigue. A complaint scale for lower respiratory tract infections is queried with the aspects of cough, mucus production, shortness of breath, sleep, ability to perform normal activities, and general feeling of illness, with gradations from 0 = normal to 6 = maximally poor. In addition, patient-reported outcomes by paper questionnaires are recorded: SF-36 V.1.0 and FACIT-F are completed in parallel to the telephone interviews from baseline to through study completion (up to 6 months); a subgroup of patients records daily changes in symptom occurrence and severity during the time of dietary supplementation (4 weeks), with gradations from 0 = not at all to 4 = intolerable.

SECONDARY OUTCOMES:
Severity of individual COVID-19 symptoms at week 0, week 2 (primary time of analysis), week 4 and week 6 as well as after 6 months. | Through study completion, up to 6 months
  Symptoms are recorded during telephone interviews at baseline, at weeks 2, 4 and 6 and after 6 months in an electronic case report form and as patient-reported outcomes by paper questionnaires (SF-36 V.1.0, FACIT-F, 4-week daily symptom questionnaire).
Frequency and severity of symptoms characteristic of post-COVID-19 syndrome (at month 6). | 6 months
  A validated smell test (Smell Identification Test™; Sensonics / MediSense) is performed by the patient and recorded as patient-reported outcome by a paper questionnaire. Questionnaires on olfactory and gustatory abilities (incl. Questionnaire of Olfactory Disorders, QOD), respiration (Multidimensional Dyspnoea Profile, MDP), mental state (Patient Health Questionnaire Depression, PHQ-8; Generalised Anxiety Disorder 7, GAD-7; Perceived Stress Scale, PSS; Brief Resilience Scale, BRS), sleep quality (Pittsburgh Sleep Quality Index, PSQI) and fatigue (Multidimensional Fatigue Inventory, MFI) are recorded as patient-reported outcomes by paper questionnaires. In addition, a cognition test (T3MS) validated for telephone interviews will be performed.
3. Levels of antibodies directed against the N protein or S protein of SARS-CoV-2 after at least 6 months (anti-S protein stratified for presence and type of booster vaccination). | 6 months
  ELISA measurements of antibodies recovered from dried blood spots are performed using a validated procedure in a central laboratory.
Frequency of complete symptom resolution after 2 weeks of dietary supplementation. | 2 weeks
  Symptoms are recorded during telephone interviews at baseline and at week 2 in an electronic case report form and as patient-reported outcomes by paper questionnaires (SF-36 V.1.0, FACIT-F, 4-week daily symptom questionnaire).
Frequency of complete symptom resolution after 4 weeks of dietary supplementation. | 4 weeks
  Symptoms are recorded during telephone interviews at baseline and at week 4 in an electronic case report form and as patient-reported outcomes by paper questionnaires (SF-36 V.1.0, FACIT-F, 4-week daily symptom questionnaire).
Frequency of complete symptom resolution after 6 weeks (4 weeks of dietary supplementation and 2 weeks follow-up). | 6 weeks
  Symptoms are recorded during telephone interviews at baseline and at week 6 in an electronic case report form and as patient-reported outcomes by paper questionnaires (SF-36 V.1.0 and FACIT-F).
Time from diagnosis resolution of individual symptoms [days]. | 6 weeks
  Symptoms are recorded during telephone interviews at baseline and at weeks 2, 4 and 6 in an electronic case report form and as patient-reported outcomes by paper questionnaires (SF-36 V.1.0, FACIT-F, 4-week daily symptom questionnaire).
Time from diagnosis to complete symptom resolution [days]. | 6 weeks
  Symptoms are recorded during telephone interviews at baseline and at weeks 2, 4 and 6 in an electronic case report form and as patient-reported outcomes by paper questionnaires (SF-36 V.1.0, FACIT-F, 4-week daily symptom questionnaire).

OTHER OUTCOMES:
World Health Organization (WHO) COVID-19 Ordinal Scale for Clinical Improvement at baseline, Week 2, Week 4 and Week 6 as well as after 6 months. | Through study completion, up to 6 months
  See https://www.who.int/publications/i/item/covid-19-therapeutic-trial-synopsis. Symptoms are recorded during telephone interviews at baseline and at weeks 2, 4 and 6 in an electronic case report form.
Frequency of severe COVID-19 (examination in an emergency department / hospitalisation with requirement for oxygen (at least 24 h), intensive care or ventilation / death by COVID-19). | Through study completion, up to 6 months
  Frequency of severe COVID-19, defined as achieving one of the following characteristics:
  1. examination in an emergency department;
  2. hospitalisation with continuous oxygen requirement of at least 24 hours;
  3. intensive care requirement;
  4. ventilation requirement;
  5. death by COVID-19.
  Characteristics are recorded during telephone interviews at baseline and at weeks 2, 4 and 6 as well as after 6 months in an electronic case report form; if necessary, the records are completed by data from the attending physicians, for which informed consent is given prior to enrolment into the trial.
Comparison between findings from the pilot phase of the study and the second part of the study. | Through study completion, up to 6 months
  Symptoms are recorded during telephone interviews at baseline and at weeks 2, 4 and 6 as well as after 6 months in an electronic case report form.
Changes in fatigue (eCRF). | Through study completion, up to 6 months
  Symptoms are recorded during telephone interviews at baseline and at weeks 2, 4 and 6 as well as after 6 months in an electronic case report form.
Changes in fatigue (FACIT-F). | Through study completion, up to 6 months
  Symptoms are recorded at baseline and at weeks 2, 4 and 6 as well as after 6 months as patient-reported outcomes by paper questionnaires (FACIT-F).
Changes in quality of life (eCRF). | Through study completion, up to 6 months
  Parameters relevant for quality of life are recorded during telephone interviews at baseline and at weeks 2, 4 and 6 as well as after 6 months in an electronic case report form.
Changes in quality of life (SF-36 V.1.0). | Through study completion, up to 6 months
  Parameters relevant for quality of life are recorded at baseline and at weeks 2, 4 and 6 as well as after 6 months as patient-reported outcomes by paper questionnaires (SF-36 V.1.0).
Changes in blood levels of tryptophan. | Through study completion, up to 6 months
  Blood levels are measured at baseline and at weeks 2, 4 and 6 as well as after 6 months (in selected patients).
Changes in blood levels of tryptophan metabolites. | Through study completion, up to 6 months
  Blood levels are measured at baseline and at weeks 2, 4 and 6 as well as after 6 months (in selected patients).
Changes in blood levels of inflammatory markers (C-reactive protein, interleukin-6, ferritin, neopterin, D-dimers). | Through study completion, up to 6 months
  Blood levels are measured at baseline and at weeks 2, 4 and 6 as well as after 6 months (in selected patients).
Changes in blood count and standard blood profile. | Through study completion, up to 6 months
  Blood count and standard blood profile are measured at baseline and at weeks 2, 4 and 6 as well as after 6 months (in selected patients).
Changes in blood metabolome composition. | Through study completion, up to 6 months
  Blood metabolome composition is measured at baseline and at weeks 2, 4 and 6 as well as after 6 months (in selected patients). Targeted metabolomics will be performed using a commercial kit for the identification of approx. 600 metabolites (MxP Quant 500, Biocrates, Innsbruck, Austria). Untargeted metabolomics will be performed by NMR.
Strain of SARS-CoV-2 virus. | 2 weeks, preferably at baseline
  Sequencing of SARS-CoV-2 virus from nasopharyngeal swab samples (in selected patients).
Changes in stool microbiome composition. | Through study completion, up to 6 months
  Stool microbiome composition is measured at baseline and at weeks 2, 4 and 6 as well as after 6 months (in selected patients). DNA will be isolated from fecal samples using DNeasy PowerSoil Kit (Qiagen), the V3-V4 region of the 16S gene amplified and barcoded amplicons will be sequenced on an Illumina MiSeq (2 x 300 nt) with >10,000 reads per sample. Reads passing quality control will be paired-end assembled and after rarefaction to normalize for sequencing depth using QIIME2 data analysis will be performed, i.e. alpha and beta diversity, taxonomic summaries, differential features, indicator analyses and correlation with metadata.
Changes in stool metagenome composition. | Through study completion, up to 6 months
  Stool metagenome composition is measured at baseline and at weeks 2, 4 and 6 as well as after 6 months (in selected patients). DNA will be isolated from fecal samples using DNeasy PowerSoil Kit (Qiagen) and sequenced on an Illumina NovaSeq 6000 using NexteraXT with 2 x 125 bp and 20x coverage. After quality filtering (removal of low-quality reads, 3' trimming, removal of reads from human DNA) MEtaGenome Analyser (MEGAN) will be used for taxonomic classification of metagenomic reads and the reads will be de novo assembled into contigs using Metagenomic Data Utilization and Analysis (MEDUSA) and then annotated to genes and functions in the Kyoto Encyclopedia of Genes and Genomes (KEGG), Clusters of Orthologous Groups (COG) and Pfam for functional analysis.
Changes in stool metabolome composition. | Through study completion, up to 6 months
  Stool metabolome composition is measured at baseline and at weeks 2, 4 and 6 as well as after 6 months (in selected patients). Targeted metabolomics will be performed using a commercial kit for the identification of approx. 600 metabolites (MxP Quant 500, Biocrates, Innsbruck, Austria). Untargeted metabolomics will be performed by NMR.
Short-term pharmacokinetics. | 3 days
  The short-term plasma pharmacokinetics after a single dose of the trial supplements (500 mg conventional nicotinamide and 500 mg nicotinamide released in a controlled manner in the intestine) will be measured in short intervals on Day 1 (every 30 min until 2 h after administration followed by hourly sampling until 12 h after administration) as well as after 24 h (Day 2) and 48 h (Day 3) in up to 5 trial participants from the subgroup of blood donors.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schreiber, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany